CLINICAL TRIAL: NCT00733564
Title: Evaluation of the Anesthetic Efficacy of Propofol,Sevoflurane and Paracervical Block for Uterine Curettage
Brief Title: Evaluation of Different Anesthesia for Uterine Curettage
Acronym: EDAUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMU-FY2008-209; NJFY0890-MZ12
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Uterine Curettage; Abortion, Induced
Keywords: Local anesthetic; Propofol; Sevoflurane
MeSH Terms: interventions — Lidocaine; Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Paracervical block will be performed
  Interventions: Drug: Lidocaine
- 2 (Experimental): Propofol anesthesia will be performed
  Interventions: Drug: Propofol
- 3 (Experimental): Sevoflurane anesthesia will be performed
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Lidocaine — Paracervical injection of 2% Lidocaine to block associated nociception input
  Other Names: Lignocaine
  Arms: 1
Drug: Propofol — Propofol 3mg/kg will be injected intravenously; 1 mg/kg will be added additionally for incomplete anesthesia
  Other Names: Diprivan
  Arms: 2
Drug: Sevoflurane — Sevoflurane 8% for anesthesia induction, 2-3% as the maintenance
  Other Names: Sevorane
  Arms: 3

SUMMARY:
Anesthesia during uterine curettage is a problem. Paracervical block is used in general for such an operation, though, the anesthetic efficacy is incomplete. Propofol is the short-lasting intravenous anesthetic administrated popularly. Sevoflurane is a new inhalational anesthetic well-known for it's "easy come, easy go" property. The investigators hypothesized that propofol, sevoflurane and paracervical block had different anesthetic efficacy during uterine curettage. Which one is the optimal selection for such operation needed to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I-II
* Performing abortion operation (medical- or surgical)
* Requiring painless abortion

Exclusion Criteria:

* < 19 yrs, and >=45 yrs
* History of central active drugs administration
* Drug abuse
* Hypertension
* Diabetes
* Any other chronic diseases
* Allergy to the study drugs
* Habit of over-volume alcohol drinking
* Records of history of centrally active drug use and psychiatry
* Any organic disorder

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Bispectral Index (BIS) value | 0, 5, 10, 20, 30min after anesthesia

SECONDARY OUTCOMES:
Intraoperative awareness | 0, 5, 10, 20, 30min after anesthesia
Vital signs | 0, 5, 10, 15, 20, 25, 30min after anesthesia
Arterial blood gas analysis | 5min before operation; 1min and 5min after beginning of the operation
Pain intensity | 0, 5, 10, 20, 30min after surgical procedures
Cortisol level | 30min before operation; 1 and 5min during operation
Side effects | 30min after operation
Uterine bleeding | 0min after completion of the operation; 1 hour after the operation

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China